CLINICAL TRIAL: NCT01608009
Title: Phase 1b Exploratory Study of [18F]Fluciclatide-PET as a Marker of Angiogenic Response to Combination Therapy With the Pan-VEGF Inhibitor, Pazopanib, and Weekly Paclitaxel in Platinum Resistant Ovarian Cancer
Brief Title: [18F]Fluciclatide-PET, Pazopanib and Paclitaxel in Ovarian Cancer
Acronym: PAZPET-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRO1627
Record Dates: First submitted 2012-03-22; First posted 2012-05-30 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Ovarian Neoplasm
Keywords: platinum resistant; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pazopanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib and paclitaxel (Experimental)
  Interventions: Drug: Pazopanib and paclitaxel

INTERVENTIONS:
Drug: Pazopanib and paclitaxel — Pazopanib 800mg od for 7 days, followed by 18 weeks of combination therapy (paclitaxel 80mg/m2 weekly and pazopanib 800mg od). Following the completion of combination therapy, patients will continue on maintenance pazopanib 800mg od until disease progression.

SUMMARY:
The purpose of this study is to assess [18F] -fluciclatide as a biomarker of response to pazopanib and to evaluate the efficacy and safety of the combination of pazopanib and paclitaxel in platinum-resistant ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of relapsed ovarian cancer
* Responded to at least on one line of prior platinum based therapy
* Relapsed within platinum resistant interval (≤6months)
* Eastern Cooperative Oncology Group (ECOG) performance status of <2
* Measurable disease defined as a lesion that can be accurately measured in at least one dimension with the longest diameter ≥25mm using conventional techniques
* Satisfactory baseline haematologic and organ function:

  * Haematologic: Absolute neutrophil count > or = 1.5 X 10^9/L; Platelets > or = 100 X 10^9/L; Haemoglobin > or = 9g/dL; PT or INR < or = 1.2 x ULN; PTT < or = 1.2 x ULN
  * Hepatic: Bilirubin < or = 1.5 X ULN; AST or ALT < or = 2.5 X ULN
  * Renal: Serum creatinine < or = 1.5 mg/dL; Or if >1.5 mg/dL, calculated creatinine clearance > or = 50mL/min; UPC <1

Exclusion Criteria:

* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg]. Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <140/90 mmHg in order for a subject to be eligible for the study.
* Treatment with any of the following anti-cancer therapies:

  * radiation therapy 28 days prior to the first dose of pazopanib OR
  * surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
  * chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
* Treatment with anti-angiogenic therapy
* Presence of gross ascites
* Clinically significant peripheral neuropathy
* Females of childbearing potential who are unwilling to avoid pregnancy, for the duration of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Assessment of change in [18F]-fluciclatide retention parameters following 1 week of pazopanib treatment | 1 week
  Semi-quantitative standardized uptake value and fully quantitative net irreversible plasma to tumour transfer constant

SECONDARY OUTCOMES:
The proportion of women who experience side effects from the combination of paclitaxel and pazopanib | 12 months
  Core study assessments including physical examination, vital signs, ECG, and adverse event reporting
The proportion of patients responding to combination paclitaxel and pazopanib | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Sharma, MD, Study Director — Imperial College London; Timothy Crook, MD, Principal Investigator — Southend University Hospital NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, London
  - Southend University Hospital NHS Foundation Trust, Southend